CLINICAL TRIAL: NCT06695403
Title: Telerehabilitation Versus Supervised Pilates Training on Exercise Capacity and Quality of Life in Lipedema Women
Brief Title: Telerehabilitation Versus Supervised Pilates Training in Lipedema Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Safaa Salem Salem Shetawy, B.Sc in Physical Therapy. Cairo University (2015). Master Degree in Physical Therapy 2021. Assistant Lecturer of Physical Therapy Suez University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012/005261
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-06

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilates Exercise (supervised versus telerehabilitation) (Experimental): 1. Pilates Exercise: The Pilates method is a low-intensity form of movement based on body control, which works the body in a complete way, promoting physical and mental health. PET is different when compared to traditional exercises, which, in turn, tend to isolate the working muscles and have specific training approaches using repetitive motions.
  2. Telerehabilitation: Telehealth is emerging as a key method for delivering essential healthcare. Primary care research suggests that telehealth is acceptable and has potential to overcome geographical barriers for individuals needing many times rehabilitation by eliminating the need for extensive and costly travel
  Interventions: Procedure: Pilates Exercise

INTERVENTIONS:
Procedure: Pilates Exercise — 1. Pilates Exercise: The Pilates method is a low-intensity form of movement based on body control, which works the body in a complete way, promoting physical and mental health. PET is different when compared to traditional exercises, which, in turn, tend to isolate the working muscles and have specific training approaches using repetitive motions.
  2. Telerehabilitation: Telehealth is emerging as a key method for delivering essential healthcare. Primary care research suggests that telehealth is acceptable and has potential to overcome geographical barriers for individuals needing many times rehabilitation by eliminating the need for extensive and costly travel
  3. Diet approach: A customized low-carbohydrate high-fat (LCHF) restricted caloric diet in women with lipedema will be used for 12 weeks. The LCHF diet may be a valuable nutritional strategy for lipedema and overweight/obese women, reducing inflammatory status with a beneficial effect on weight, glucose profile the concentration of

SUMMARY:
1. Pilates Exercise: The Pilates method is a low-intensity form of movement based on body control, which works the body in a complete way, promoting physical and mental health. PET is different when compared to traditional exercises, which, in turn, tend to isolate the working muscles and have specific training approaches using repetitive motions.
2. Telerehabilitation: Telehealth is emerging as a key method for delivering essential healthcare. Primary care research suggests that telehealth is acceptable and has potential to overcome geographical barriers for individuals needing many times rehabilitation by eliminating the need for extensive and costly travel
3. Diet approach: A customized low-carbohydrate high-fat (LCHF) restricted caloric diet in women with lipedema will be used for 12 weeks. The LCHF diet may be a valuable nutritional strategy for lipedema and overweight/obese women, reducing inflammatory status with a beneficial effect on weight, glucose profile the concentration of triglycerides and HDL

ELIGIBILITY:
Inclusion Criteria:

1. Sixty female patients diagnosed with lipedema.
2. Their ages will range from 35-45 years old.
3. Patients diagnosed with lipedema ≥ 5 years.
4. Patients with grade 2 and 3 lipedema.
5. Patients with type 2 and 3 lipedema.
6. Patients with BMI ≥ 25 kg/m2
7. All patients will be clinically stable.

Exclusion Criteria:

Patient with any of the following will be excluded from the study:

1. Patients with lower limb edematous diseases such as lymphedema or chronic venous insufficiency.
2. Patients with history of previous liposuction.
3. Patients with asymmetrical lower limbs.
4. Patients with history of bariatric surgeries.
5. Patients on weight loss medications.
6. Patients any medical condition prohibiting exercise (cardiac pacemakers, diabetes mellitus, uncontrolled hypertension, and congestive heart failure)
7. Pregnant females.
8. Patients with BMI ≥ 40 kg/m2 (morbid obese).
9. Cancer patients (patients on chemotherapy, immunotherapy radiopathy).
10. Infectious diseases (HIV/AIDS, HCV, and Tuberculosis).
11. Chronic inflammatory autoimmune disease such as Sjogren's syndrome
12. Patients with neurological disorders: stroke and epilepsy.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females who have lipedema
Enrollment: 60 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Six minutes walk test | 12 weeks
  Procedures for the 6MWT will be adopted from the American Thoracic Society (ATS) guidelines . 6MWT is used to assess exercise tolerance
World Health Organization's Quality of Life questionnaire (WHOQOL BREF): | 12 weeks
  The World Health Organization (WHO) has defined "QOL" as "an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns". Recently, many general instruments have been used to measure QOL in different groups (e.g., patients, workers, population and so on). One of these instruments is the World Health Organization QOL-BREF (WHOQOL-BREF) questionnaire which captures many subjective aspects of QOL
Limb Circumference | 12 weeks
  Limb Circumference: These measurements of definite points diameter in lower extremities using tape measurement are also used to predict progression and as follow up instrument

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes